CLINICAL TRIAL: NCT00521053
Title: A Phase 2 Study of Intralesional PV-10 in the Treatment of Metastatic Melanoma
Brief Title: Phase 2 Study of Intralesional PV-10 for Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Provectus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PV-10-MM-02
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Results first posted 2014-08-25 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Melanoma
Keywords: immune; vaccine; systemic; Metastatic Melanoma (AJCC Stage III or IV)
MeSH Terms: conditions — Melanoma | interventions — Rose Bengal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PV-10 (Experimental)
  Interventions: Drug: PV-10 (10% rose bengal disodium)

INTERVENTIONS:
Drug: PV-10 (10% rose bengal disodium) — Intralesional injection for chemoablation

SUMMARY:
The primary objective of this study is to investigate the effectiveness of intralesional (IL) PV-10 for locoregional treatment of metastatic melanoma. This study will also include assessment of response in untreated bystander lesions following intralesional injection of PV-10 into targeted lesions. Additional objectives are to determine the safety profile of PV-10 following intralesional injection, and assess the pharmacokinetic profile of PV-10 in the bloodstream following intralesional injection.

DETAILED DESCRIPTION:
This is a multicenter, open-label, single-agent study. Subjects with at least one melanoma lesion ≥ 0.2 cm in diameter that can be accurately measured by ruler/caliper or ultrasound will receive intralesional injection of PV-10 into each of up to twenty (20) Study Lesions. Additionally, one to two measurable Bystander Lesions may remain untreated and will be followed for assessment of bystander response.

To accurately reflect anticipated clinical use, repeat dosing of treated lesions will be allowed at the Investigator's discretion at weeks 8, 12 and 16 following initial treatment for those lesions not exhibiting complete response. Subjects will be followed for 52 weeks following initial treatment with PV-10.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, age 18 years or older.
* Histologically or cytologically confirmed metastatic melanoma, AJCC (2002) Stage III (regional lymph node metastasis, in-transit metastasis or satellite metastasis) or Stage IV (distant metastasis).
* Measurable disease in at least one lesion ≥ 0.2 cm in diameter that can be accurately measured by ruler/caliper or ultrasound. Target, Non-Target and Bystander Lesions selected by discretion of Investigator.
* Performance Status: ECOG 0-2.
* Life Expectancy: At least 6 months.
* Hematopoietic:

  * White blood cell count (WBC) no less than 2500/mm3 (2.5 x 10E9/L).
  * Absolute neutrophil count (ANC) no less than 1,000/mm3 (1.0 x 10E9/L).
  * Platelet count no less than 90,000/mm3 (90 x 10E9/L).
* Blood Chemistry:

  * Creatinine no greater than 1.5 times the upper limit of normal (ULN).
  * Total bilirubin no greater than 1.5 times the upper limit of normal (ULN).
  * AST/ALT no greater than 3 times the upper limit of normal (ULN).
* Thyroid Function:

  * Total T3 or free T3 (serum triiodothyronine), total T4 or free T4 (serum thyroxine) and THS (serum thyrotropin) within normal limits.
* Cardiovascular Function:

  * No clinically significant cardiovascular disease.
* Respiratory Function:

  * No clinically significant respiratory disease.
* Immunological Function:

  * No known immunodeficiency disease. Subjects must have adequate immune system function in the opinion of the Investigator.

Exclusion Criteria:

* Radiation therapy within 4 weeks of study treatment or to any Study Lesion within 12 weeks of study treatment.
* Chemotherapy:

  * Chemotherapy or other systemic cancer therapy within 4 weeks of study treatment (6 weeks for nitrosoureas or mitomycin).
  * Regional chemotherapy (limb infusion or perfusion) within 12 weeks of study treatment.
* Local treatment (e.g., surgery, cryotherapy, radiofrequency ablation) to the treatment area within 4 weeks of study treatment.
* Investigational agents within 4 weeks (or 5 half-lives) of study treatment.
* Photosensitizing agents within 5 half-lives of study treatment.
* Anti-tumor vaccine therapy within 6 weeks of study treatment.
* Concurrent or Intercurrent Illness:

  * Severe diabetes.
  * Extremity complications due to diabetes.
  * Significant concurrent or intercurrent illness, psychiatric disorders, or alcohol or chemical dependence that would, in the opinion of the Investigator, compromise their safety or compliance or interfere with interpretation of study results.
  * Thyroid disease (subclinical or ongoing), goiter, partial thyroidectomy, previous radioiodine- or surgically-treated Graves' hyperthyroidism or cystic fibrosis, or taking thyroid hormone medication.
* Pregnancy:

  * Female subjects who are pregnant or lactating.
  * Female subjects who have positive serum ßHCG pregnancy test taken within 7 days of PV-10 treatment.
  * Fertile subjects who are not using effective contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-09; Primary Completion 2010-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John F Thompson, MD, Principal Investigator — Sydney Melanoma Unit
Locations (7):
- United States (4):
  - California Pacific Medical Center, San Francisco, California
  - University of Louisville, Louisville, Kentucky
  - St Luke's Hospital & Health Network, Bethlehem, Pennsylvania
  - M.D. Anderson Cancer Center, Houston, Texas
- Australia (3):
  - Sydney Melanoma Unit, Sydney, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia

RESULTS

PARTICIPANT FLOW:
Groups:
- PV-10: PV-10 (10% rose bengal disodium): Intralesional injection for chemoablation. In the treatment phase, participants received a single IL injection of PV-10 into each of up to 20 study lesions on day 0 (i.e., one cycle). Treatment cycles could be repeated at weeks 8, 12 and 16 for new non-target lesions or existing target or non-target lesions not exhibiting complete response (i.e., complete disappearance). Participants were observed for 52 weeks. Radiologic assessments of visceral disease status were performed every 12 weeks throughout the study and patients were transitioned into survival follow-up if at any time the investigator identified clinical or radiologic evidence of distant progression. No other melanoma therapy was permitted during the study interval.
Period: Treatment Phase
Arm/Group | PV-10
Started | 80
Received 1 Cycle of PV-10 | 35
Received 2 Cycles of PV-10 | 26
Received 3 Cycles of PV-10 | 16
Received 4 Cycles of PV-10 | 3
Completed | 80
Not Completed | 0
Period: Observation Phase
Arm/Group | PV-10
Started | 80
Completed | 12
Not Completed | 68
Not completed — Disease Progression | 55
Not completed — Additional PV-10 via alternate protocol | 8
Not completed — Death | 2
Not completed — Adverse Event | 1
Not completed — Other non-study melanoma treatment | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | PV-10
Number analyzed (Participants) | 80
Age, Continuous [Median (Full Range); unit: years] | 70.0 [33 to 97]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 48
Region of Enrollment [Number; unit: participants]
  United States | 27
  Australia | 53
American Joint Committee on Cancer (AJCC) Stage at Baseline [Number; unit: participants] — Participants were staged clinically at baseline based on cutaneous and subcutaneous, nodal and visceral tumor burden. Stage III participants had disease confined to cutaneous, subcutaneous and/or nodal sites. Stage IV participants had distant metastatic disease (i.e., distant cutaneous or subcutaneous metastases or visceral metastases).
  participants
    IIIB | 38
    IIIC | 24
    M1a | 3
    M1b | 5
    M1c | 10
Tumor Burden in Skin [Number; unit: participants]
  Less than 10 Lesions | 44
  10 or more Lesions | 29
  Too Numerous to Count | 7
Prior Interventions [Number; unit: participants] — Participants may have had more than one prior intervention.
  participants
    Excision | 80
    Nodal Biopsy | 50
    Regional Chemotherapy | 19
    Immunotherapy | 17
    Radiotherapy | 17
    Investigational Agents | 11
    Systemic Chemotherapy | 10
    Distal Amputation | 7
    Other | 6
Number of Prior Interventions [Median (Full Range); unit: prior interventions] | 6 [1 to 19]
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Participants were staged clinically at baseline using the ECOG Performance Status scale:
  GRADE 0: Fully active, able to carry on all pre-disease performance without restriction. GRADE 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work. GRADEe 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours.
  participants
    0 | 53
    1 | 25
    2 | 2
Untreated Disease Burden [Number; unit: participants] — Participants were categorized at baseline according to tumor burden that was not injected with PV-10.
  participants
    Untreated Visceral Disease | 18
    One or More Lesions Not Measured and Untreated | 8
    All Lesions Treated Except Bystanders | 26
    All Lesions Treated | 28

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) of PV-10 Treated Lesions
Description: Using modified Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for cutaneous or subcutaneous target lesions assessed by ruler, caliper or ultrasound: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response Rate (ORR) = %CR + %PR.
Time Frame: 52 weeks
Population: ITT participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PV-10
Number analyzed (Participants) | 80
percentage of participants | 51.3 [39.8 to 62.6]

2. Secondary Outcome: Objective Response Rate of Untreated Bystander Lesions
Description: Using modified Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for designated, untreated cutaneous or subcutaneous bystander lesions assessed by ruler, caliper or ultrasound: Complete Response (CR), disappearance of all bystander lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of bystander lesions; Objective Response Rate (ORR) = %CR + %PR.
Time Frame: 52 weeks
Population: ITT participants having at least one uninjected dermal bystander lesion designated at baseline (some ITT participants did not have at least one bystander lesion).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PV-10
Number analyzed (Participants) | 42
percentage of participants | 33.3 [19.6 to 49.6]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression is defined using modified Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or significant worsening of non-target disease (e.g., a measurable increase in non-target lesions or the appearance of new lesions) indicative of disease progression.
Time Frame: 52 weeks
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Stage III: Participants reporting Stage III disease at baseline
- Stage IV: Participants reporting Stage IV disease at baseline
Arm/Group | Stage III | Stage IV
Number analyzed (Participants) | 62 | 18
Months | 3.7 [2.9 to 4.5] | 1.9 [1.6 to 2.1]

4. Post Hoc Outcome: Rate of Complete Response
Description: Using modified Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for cutaneous or subcutaneous target lesions assessed by ruler, caliper or ultrasound: Complete Response (CR), disappearance of all target lesions; Complete Response Rate (CRR) = %CR.
Time Frame: 52 weeks
Population: ITT participants having all baseline disease injected with PV-10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Lesions Treated
Number analyzed (Participants) | 28
percentage of participants | 50 [30.6 to 69.4]

5. Secondary Outcome: Overall Survival
Description: 1-year survival
Time Frame: 52 weeks
Population: ITT participants
Measure: Number; unit: percentage of participants
Arm/Group | Stage III | Stage IV
Number analyzed (Participants) | 62 | 18
percentage of participants | 89 [1.25 to 13.38] | 39

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the study interval (52 weeks) and followed until resolution. Events on-going at time of withdrawal were followed until resolution or for a period of at least 28 days from last dose of study medication.
Arm/Group | PV-10
Serious Adverse Events (participants affected / at risk) | 14/80
Other Adverse Events (participants affected / at risk) | 80/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PV-10 (N=80)
Left ventricular hypertrophy (Cardiac disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Injection site oedema (General disorders) | 1
Injection site swelling (General disorders) | 2
Injection site ulcer (General disorders) | 1
Pyrexia (General disorders) | 1
Viral infection (Infections and infestations) | 1
Injection site necrosis (General disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Pneumonia (Infections and infestations) | 2
Back injury (Injury, poisoning and procedural complications) | 1
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 1
Injection site pain (General disorders) | 2
Injection site infection (General disorders) | 1
Injection site vesicles (General disorders) | 1
Pituitary disorder (Endocrine disorders) | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PV-10 (N=80)
Abdominal pain (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 10
Diarrhoea (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 17
Vomiting (Gastrointestinal disorders) | 7
Fatigue (General disorders) | 5
Injection site cellulitis (General disorders) | 4
Injection site discolouration (General disorders) | 25
Injection site erythema (General disorders) | 11
Injection site infection (General disorders) | 5
Injection site inflammation (General disorders) | 6
Injection site oedema (General disorders) | 32
Injection site pain (General disorders) | 65
Injection site photosensitivity reaction (General disorders) | 6
Injection site pruritus (General disorders) | 17
Injection site rash (General disorders) | 4
Injection site swelling (General disorders) | 20
Injection site ulcer (General disorders) | 4
Injection site vesicles (General disorders) | 30
Injection site warmth (General disorders) | 4
Lethargy (General disorders) | 4
Oedema peripheral (General disorders) | 5
Nasopharyngitis (Infections and infestations) | 6
Decreased appetite (Metabolism and nutrition disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5
Headache (Nervous system disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less